CLINICAL TRIAL: NCT07300995
Title: A Behavioral Pain Intervention for Older Breast Cancer Patients in Medically Underserved Areas
Brief Title: Behavioral Pain Intervention for Older Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00117948; P30AG022845 (NIH)
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: cancer; pain; coping; symptom management
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Coping Skills Training (Experimental): Participants in this group will complete a 50-minute telehealth session with a trained study nurse. During this session, they will be taught how to use several coping strategies for managing pain. This will be followed by 5 weekly, 15-minute supportive phone calls, where the study nurse will reinforce the learned coping skills. They will be asked to complete 2 follow-up surveys (10 weeks and 15 weeks after the first survey).
  Interventions: Behavioral: Pain Coping Skills Training (PCST)
- Usual Care (No Intervention): Participants in this group will not complete the new program. They will be asked to complete 2 follow-up surveys (10 and 15 weeks after the first survey).

INTERVENTIONS:
Behavioral: Pain Coping Skills Training (PCST) — Behavioral pain intervention delivered via telehealth.
  Arms: Pain Coping Skills Training

SUMMARY:
This randomized controlled trial examines a 1-session, telehealth pain coping skills training (PCST) protocol with five 15-minute maintenance calls (Brief PCST-Community) adapted for women with breast cancer in medically underserved areas. Pain, health-related quality of life, and self-efficacy for pain management will be assessed at baseline and 10 and 15 weeks later.

DETAILED DESCRIPTION:
Pain continues to be persistent, interfering, and distressing for women with breast cancer. Behavioral cancer pain interventions continue to be poorly implemented with pronounced disparities for older breast cancer patients receiving oncology care in medically underserved areas. Within this context, this randomized controlled trial examines a 1-session, telehealth pain coping skills training (PCST) protocol with five 15-minute maintenance calls (Brief PCST-Community) adapted for women with breast cancer in medically underserved areas. Pain, health-related quality of life, and self-efficacy for pain management will be assessed at baseline and 10 and 15 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Receiving cancer care at a Duke Cancer Network (DCN) clinic
* Stage I-IV breast cancer
* Self-reported pain on at least 10 days in the last month and pain rating of worst pain of 4 or greater on a 0-10 scale in the last week
* Biologically female
* Greater than or equal to 55 years old
* Ability to speak and read English
* Hearing and vision that allows for successful completion of videoconferencing and phone session

Exclusion Criteria:

* Participation in the last 6 months in a pain coping skills training program

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain severity as measured by the Brief Pain Inventory (BPI) | Baseline, 10-week assessment, 15-week assessment
  BPI Pain Severity (worst, least, average, current pain on 0-10 scale) scores are averaged for a total score range of 0 to 10, with higher scores indicating greater pain severity.
Pain interference as measured by the Brief Pain Inventory (BPI) | Baseline, 10-week assessment, 15-week assessment
  BPI Pain Interference (7 daily life areas such as mood, sleep, activity rated 0-10) scores are averaged for a total score range of 0 to 10, with higher scores indicating greater pain interference.
Health Related Quality of Life (HR-QOL) as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) - Physical Function | Baseline, 10-week assessment, 15-week assessment
  A PROMIS Physical Function T-score is a standardized number (mean 50, SD 10) from the Patient-Reported Outcomes Measurement Information System (PROMIS) that reflects self-reported physical ability with higher scores indicating better function.
Health Related Quality of Life (HR-QOL) as measured by the Patient Reported Outcomes Measurement Information System (PROMIS-29) - Mental Health | Baseline, 10-week assessment, 15-week assessment
  A PROMIS Mental Health T-score is a standardized number (mean 50, SD 10) from the Patient-Reported Outcomes Measurement Information System (PROMIS) that reflects self-reported mental health with higher scores indicating worse mental health.

SECONDARY OUTCOMES:
Self-Efficacy for Pain Management | Baseline, 10-week assessment, 15-week assessment
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item scale rating confidence (0-6) in specific tasks despite pain. The total score ranges from 0 to 60, where higher scores indicate greater self-efficacy.

IPD SHARING:
Plan to Share IPD: No